CLINICAL TRIAL: NCT02865057
Title: Ultrasound Examination as a Teaching Tool for Vaginal Exam Assessment of Fetal Position in Active Labor
Brief Title: Assessment of Fetal Position in Active Labor
Acronym: U/S
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MFM Fellow, St. Louis University
Other Study IDs: 26057
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3rd year Residents: 3rd year Ob, Gyn Residents
  Interventions: Procedure: Vaginal assessment
- 4th Year Residents: 4th year Ob, Gyn Residents
  Interventions: Procedure: Vaginal assessment

INTERVENTIONS:
Procedure: Vaginal assessment — Vaginal assessment of position prior to delivery

SUMMARY:
Vaginal exams are used routinely in labor to assess cervical dilation and position of the baby (facing anterior, facing to the right or left side, facing towards maternal spine). This technique has a widely variable accuracy rate (24.0-85.6%). Ultrasound has been used to help confirm or correct the vaginal assessment by obstetricians, but has not been used to assess the utility of immediate feedback to improve the accuracy of vaginal assessment by physicians in training. The investigators plan to use ultrasound assessment to determine if this education is effective in increasing accuracy in the resident population.

DETAILED DESCRIPTION:
Residents will be informed of the study through an education session (as a group) and then be consented individually. Each resident will complete 15 baseline exams, 20 exams with immediate ultrasound confirmation, and 15 exams for post-test baseline. Exams will take place periodically throughout the year. Both 3rd and 4th year residents will be assessed during the same time period by the MFM fellows. Ultrasounds will follow the vaginal exam as closely as possible to prepare for delivery. A picture of the fetal position (with no name or MRN) for documentation to be taken during the SOC ultrasound and kept in the research chart for the resident.

In training feedback is not always standard. This teaching tool, consistent and standard feedback with regard to the correlation between vaginal exam and ultrasound, would allow the resident to learn to assess fetal position more accurately.

Information from the maternal chart (history and delivery information) will be collected as de identified. Data will be recorded on the data collection sheet which is labeled with a code number linking the resident participant only.

Data collected from the residents will be assigned a random Code numbers used to link the subject to their data.

Code and identifiers will be kept separate. Paper copies will be kept in a locked cabinet, in a locked office, in a locked suite.

ELIGIBILITY:
Inclusion Criteria:

* Physicians in obstetrics training -

Exclusion Criteria:

* Physicians outside of obstetrics training.

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 3rd and 4th year Ob, Gyn Residents
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
assessing fetal position | Immediate
  Categorical variables will be expressed as frequencies and percentages. Continuous variables will be expressed as means and standard deviations and/or medians and ranges. Demographic characteristics will be assessed using chi-square test and Fischer's Exact test for categorical variables. To examine improvement in the number of correct physical exams from baseline to post-intervention a repeated measures t-test or Wilcoxon signed rank test will be performed. An independent measures t-test or Mann-Whitney U test will be performed to compare the number of correct physical exams between resident groups. Other pertinent statistical tests will be utilized as needed to account for group differences and control for variables of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No